CLINICAL TRIAL: NCT02626468
Title: Validation in Healthy Subjects and Different Diagnostic States
Brief Title: Validation of Structured Light Plethysmography - Health and Disease
Acronym: SLP-RespDis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pneumacare Ltd (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PMC-T3D-004
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Participants with no diagnosis of respiratory disease between the ages of 0 and 80
- COPD: Patients from different diagnostic groups between the ages of 0 and 80

SUMMARY:
Validation of Structured Light Plethysmography (SLP) in patients with conditions such as Chronic Obstructive Pulmonary Disease (COPD) that effect breathing and in healthy participants.

DETAILED DESCRIPTION:
The investigators hypothesize that SLP may be a useful tool to differentiate between different respiratory diseases. To further examine differences in disease and health, and between diseases SLP measurements will be recorded in a range of diagnostic conditions that effect breathing and in healthy normal subjects.

This is a non-randomised observational study to validate Structured Light Plethysmography in two groups of participants: those with Respiratory condition such as COPD and a normal healthy group. Neither group will receive any clinical intervention. SLP data capture and spirometry (as part of the patients clinical care) will be performed by the patients. The data collected from this study will allow examination of different breathing patterns between patients with different diseases, to compare breathing patterns in patients to those in healthy individuals, and to compare breathing patterns within a healthy population.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 0 and 80 years

Exclusion Criteria:

* Any contraindication to spirometry (if performed) or a history of a myocardial infarction or chest surgery within 4 weeks
* Patient unable to sit in an upright (or supine in the case of infants) position for required period of time
* Patients with significant co morbidities (assessed by the clinician at screening only):
* Chest wall or spinal deformity e.g. scoliosis
* Obstructive Sleep Apnoea (OSA) Apnoea hypopnoea index > 30 (if known)
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in the study
* BMI > 40
* Inability to consent/comply with trial protocol

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A range of diagnostic conditions that effect breathing and healthy normal subjects. The study will aim to recruit:
  200 patients from different diagnostic groups between the ages of 0 and 80 100 healthy participants with no diagnosis of respiratory disease, between the ages of 0 and 80
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Difference in SLP Breath Timing indices and measured in seconds and between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing
Difference in SLP Breath Timing Ratios between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the trace of movement over time of the thoracoabdominal (TA) wall during tidal breathing
Difference in SLP derived Relative Contribution (measured in %) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing that describes the contribution of a region of the thoracoabdominal wall to total displacement
Difference in SLP derived Phase (measured in degrees) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the movement of the thoracoabdominal (TA) wall during tidal breathing that describes the contribution of a region of the thoracoabdominal wall to total displacement
Difference in SLP derived displacement rate derived parameters (measured in distance per second) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters derived from the trace of displacement rate over time of the thoracoabdominal (TA) wall during tidal breathing
Difference in SLP displacement rate derived ratios between Patients and Healthy Subjects (measured in distance per second) between Patients and Healthy Subjects | Baseline
  SLP breathing parameters ratios derived from the trace of displacement rate over time of the thoracoabdominal (TA) wall during tidal breathing

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | Baseline
  Measurement of FEV1
Forced Vital Capacity (FVC) | Baseline
  Measurement of FVC

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] de Boer WH, Lasenby J, Cameron J, Wareham R, Ahmad S, Roach C, Hills W, Iles R. SLP: a zero-contact non-invasive method for pulmonary function testing. In: Labrosse F, Zwiggelaar R, Liu Y, Tiddeman B, eds, Proceedings of the British Machine Vision Conference. BMVA Press, 2010; pp 85.1-85.12
- [Background] Morgan MD, Gourlay AR, Denison DM. An optical method of studying the shape and movement of the chest wall in recumbent patients. Thorax. 1984 Feb;39(2):101-6. doi: 10.1136/thx.39.2.101. PMID 6701820